CLINICAL TRIAL: NCT04891861
Title: A Pilot Trial of Restarting Direct Oral Anticoagulants After Traumatic Intracranial Hemorrhage
Brief Title: Restart TICrH Alpha Pilot Protocol, Restarting DOACs After Traumatic Intracranial Hemorrhage
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Texas at Austin (Other)
Collaborators: University of Kansas (Other)
Responsible Party: Principal Investigator, Truman J Milling Jr, Research Director SDMS Stroke Institute, University of Texas at Austin
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ML42205
Record Dates: First submitted 2021-05-10; First posted 2021-05-19 (Actual); Last update posted 2021-05-19 (Actual); Status verified 2021-05

CONDITIONS: Anticoagulants; Increased
Keywords: restart; anticoagulant; DOAC
MeSH Terms: interventions — apixaban; Rivaroxaban; edoxaban; Dabigatran

STUDY DESIGN:
Intervention Model Description: Randomized trial of 1 versus 4 week DOAC restart after TICrH
Who Masked: Outcomes Assessor
Masking Description: Central blinded assessment of endpoints
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1 week restart (Active Comparator): restart DOAC at 1 week post injury at label dose and frequency
  Interventions: Drug: Apixaban
- 4 week restart (Active Comparator): restart DOAC at 4 weeks post injury at label dose and frequency
  Interventions: Drug: Apixaban

INTERVENTIONS:
Drug: Apixaban — Direct Oral Anticoagulation all at label dose and frequency
  Other Names: Rivaroxaban; Edoxaban; Dabigatran

SUMMARY:
Randomized pilot trial of restarting DOACs at 1 week versus 4 weeks after traumatic intracranial hemorrhage

DETAILED DESCRIPTION:
Restart TICrH two-center pilot trial will assign patients with anticoagulant-associated traumatic intracranial hemorrhage to restart anticoagulation at 1 week or 4 weeks. Entry into the trial is primarily driven pragmatically by clinician intent to restart any Direct Oral Anticoagulant (DOAC, i.e. apixaban, rivaroxaban, edoxaban, dabigatran. There is no head to head evidence of superiority of any drug) after anticoagulant-associated traumatic intracranial hemorrhage and equipoise concerning restart of anticoagulation at the specified time intervals. DOAC will be at label dose with label adjustments for creatinine clearance. DOAC will be at continuation dose, i.e. not initial therapy high doses in the setting of VTE.

ELIGIBILITY:
Inclusion Criteria:

1. Acute traumatic intracranial hemorrhage on anticoagulation for Atrial Fibrillation (AF) or Venous Thromboembolism (VTE)
2. Patient is higher risk for stroke or other thrombotic events as witnessed by having a CHA2DS2-VASc score of > 3 (at least 3 of the following risk factors: age greater than 65, (age > 75 counts for 2 points), history of stroke or TIA (2 points), history of heart failure, history of diabetes, history of atherosclerotic vascular disease, female biological sex, history of hypertension)
3. DOAC prescribed at label dose with creatinine clearance adjustments. DOAC at continuation dose, i.e., not initial therapy high doses in the setting of VTE

Exclusion Criteria:

1. Mechanical Valve or Ventricular Assist Device (VAD)
2. SDH >8 mm maximum width or any midline shift at any time point or more than one SDH
3. Physician plan to start/restart antiplatelet therapy during trial period
4. Abbreviated Injury Scale other than head >3
5. Pregnancy
6. Inability to understand need for adherence to study protocol
7. Renal function below DOAC label exclusions
8. Any active pathological bleeding (e.g. no acute blood on most recent CT)
9. Hypersensitivity to drug or other label contraindication
10. Any bleeding that the investigator deems unsafe to restart DOAC at 1 week post injury, or conversely unsafe to hold DOAC to 4 weeks
11. Completion of DOAC therapy expected prior to 60 day primary endpoint, e.g. 3-6 month VTE treatment
12. Concomitant need for strong inducers/inhibitors of p-gp and CYP3A4
13. Low body weight (<45kg)
14. Inability to swallow

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-07-01 (Estimated); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
60-day composite endpoint | 60 days
  A 60-day composite endpoint that includes the following clinical events: New or expansion of intracranial hemorrhage, other BARC3a or above major hemorrhage 28, stroke, systemic embolism, myocardial infarction, proximal lower extremity deep vein thrombosis, pulmonary embolism and cardiovascular death

SECONDARY OUTCOMES:
Disability Rating Scale (0-29 scale range) | 60 days
  Functional Measure
Modified Rankin Scale (0-6 scale range) | 60 day
  Functional Measure
Standard Gamble | pre-randomization (The day before randomization, which must occur within 6 days of index injury) and after endpoints (the day after one of the endpoints occurs. We cannot know precisely when this will occur in the 60 day follow up period)
  The standard gamble is the gold standard for analysis of decision making under uncertainty 7. It is an interview technique that begins with a description of a disease state. The patient is then asked to imagine suffering the disease and having a choice between taking a medication that might cure them but also might kill them. The so-called ping-pong method requires the interviewer to start with a hypothetical scenario of 0% probability of cure and 100% probability of a painless instant death. The interviewer then asks the patient if they would take the medication. He then flips the scenario, 100% cure, 0% death. He then goes back and forth between successive scenarios of lower death higher cure and lower cure higher death. Eventually, the patient settles at an equipoise and indecision of whether the risk of dying is worth incurring to take the medication and cure the disease. This is the patient's utility for that disease, expressed as a number between 0 and 1.

IPD SHARING:
Plan to Share IPD: Yes
Sharing via BIOLINCC
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After primary publication

REFERENCES:
- [Result] Milling TJ Jr, Warach S, Johnston SC, Gajewski B, Costantini T, Price M, Wick J, Roward S, Mudaranthakam D, Dula AN, King B, Muddiman A, Lip GYH. Restart TICrH: An Adaptive Randomized Trial of Time Intervals to Restart Direct Oral Anticoagulants after Traumatic Intracranial Hemorrhage. J Neurotrauma. 2021 Jun 1;38(13):1791-1798. doi: 10.1089/neu.2020.7535. Epub 2021 Apr 6. PMID 33470152